CLINICAL TRIAL: NCT04665206
Title: Phase I/II, Multi-Center, Open-Label Study of VT3989, Alone or in Combination, in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study to Evaluate VT3989 in Patients With Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vivace Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VT3989-001
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor, Adult; Mesothelioma; NSCLC
MeSH Terms: conditions — Mesothelioma | interventions — Nivolumab; Ipilimumab; osimertinib

STUDY DESIGN:
Intervention Model Description: Part 1 dose escalation: 3 + 3 design Part 2 dose expansion: up to 6 cohorts Part 3 combination: 2 cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VT3989 Dose Escalation [Not Recruiting] (Experimental): VT3989 dosed orally in 21 or 28 day cycles. Patients will be enrolled into escalating dose levels during the Dose Escalation Phase
  Interventions: Drug: VT3989
- Dose Expansion [Not Recruiting] (Experimental): VT3989 dosed in 21 or 28 day cycles in patients with refractory metastatic solid tumors or mesothelioma.
  Interventions: Drug: VT3989
- Combination [Recruiting] (Experimental): VT3989 dosed in 28 day cycles in patients with metastatic solid tumors or mesothelioma, in combination with immunotherapy (nivolumab/ipilimumab) or targeted therapy (osimertinib)
  Interventions: Drug: VT3989; Drug: Nivolumab & Ipilimumab; Drug: Osimertinib

INTERVENTIONS:
Drug: VT3989 — 25, 50, 100, 150 or 200 mg capsules for oral administration.
Drug: Nivolumab & Ipilimumab — Nivolumab infusion - 360 mg every 3 weeks, 30-minute intravenous infusion
  Ipilimumab infusion - 1 mg/kg every 6 weeks, 30-minute intravenous infusion
  Arms: Combination [Recruiting]
Drug: Osimertinib — 40 or 80 mg tablets for oral administration
  Arms: Combination [Recruiting]

SUMMARY:
This is an open-label, dose escalation and expansion study to evaluate the safety, tolerability, PK, and biological activity of VT3989 administered, alone or in combination, once daily in patients with mesothelioma and/or metastatic solid tumors that are resistant to standard therapy or for which no effective standard therapy is available.

DETAILED DESCRIPTION:
Dose escalation (Part 1) will employ a traditional 3 + 3 design to assess safety of VT3989 in patients with metastatic solid tumors or mesothelioma. The 3 + 3 design will be implemented until the MTD or recommended phase 2 dose(s) and schedule(s) are determined. The MTD is defined as the highest dose level at which < 33% of patients experience a dose limiting toxicity (DLT) during the first cycle of the study (Cycle 1).

Dose Expansion (Part 2) will further evaluate the safety and assess preliminary antitumor activity at the recommended phase 2 dose(s) and schedule(s) with up to 6 cohorts. Expansion cohorts 1 and 2 will enroll patients with mesothelioma of any site origin with or without NF2 mutations. Expansion cohort 3 will enroll non-pleural mesothelioma patients. Expansion cohort 4 will enroll solid tumor patients with clearly inactivating NF2 mutations/alterations or YAP/TAZ gene rearrangements. Cohort 5 will enroll pleural mesothelioma patients.

Combination part (Part 3) includes two cohorts. Cohort A will enroll mesothelioma patients who will receive VT3989 in combination with immunotherapy (nivolumab plus ipilimumab). Cohort B will enroll NSCLC patients whose tumors have exon 19 deletion or exon 21 L858R mutation and will receive VT3989 in combination with targeted therapy (Osimertinib).

ELIGIBILITY:
Inclusion Criteria:

* Part 3 Combination Cohort A: Patients with pathologically diagnosed, metastatic or unresectable malignant mesothelioma (including both pleural and non-pleural) who have not received systemic therapy.
* Part 3 Combination Cohort B: Patients with pathologically diagnosed incurable locally advanced (inoperable or recurrent), or metastatic NSCLC with exon 19 deletions or exon 21 L858R mutations, with or without prior treatment with Osimertinib.
* Measurable disease per RECIST v1.1 for non-pleural mesothelioma or other solid tumors or modified RECIST v1.1 for malignant pleural mesothelioma. mRECIST may be used for pleural extension of non-pleural mesothelioma or for mixed pleural and peritoneal (or other) mesothelioma.
* ECOG: 0-1.
* Adequate organ functions, including the liver, kidneys, and hematopoietic system.

Exclusion Criteria:

* Active brain metastases or primary CNS (central nervous system) tumors.
* History of leptomeningeal metastases
* Active or chronic, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Known HIV positive or active Hepatitis B or Hepatitis C
* Clinically significant cardiovascular disease
* Corrected QT (QTcF) interval > 470 msec (using Fridericia's correction formula); except for Part 2 Expansion Cohort 3, the QTcF interval criteria is > 450 msec).
* Additional active malignancy that may confound the assessment of the study endpoints
* Women who are pregnant or breastfeeding
* Prior treatment with TEAD inhibitor, except for EHE patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity | over the first 21 days of dosing
  Incidence of Adverse and Serious Adverse Events
Occurrence of General Toxicity | through study completion, an average of 30 months
  Incidence of Adverse and Serious Adverse Events, Discontinuations due to Adverse Events and general safety evaluations

SECONDARY OUTCOMES:
Tumor Response | through study completion, an average of 30 months
  Determined by RECIST v1.1 or modified RECIST v1.1
Pharmacokinetic Evaluation - Cmax | for first 6 cycles
  Peak plasma concentration of VT3989
Pharmacokinetic Evaluation - Tmax | for first 6 cycles
  Time to reach peak plasma concentration of VT3989
Pharmacokinetic Evaluation - Half-life | for first 6 cycles
  Time required for the plasma concentration of VT3989 to reduce by half after reaching peak
Overall survival (Part 2, expansion cohort 3, 4, and 5) | Through study completion, an average of 30 months
  The overall survival of the enrolled patients from starting VT3989 treatment
Progression free survival (Part 2, expansion cohort 3, 4, and 5) | Through study completion, an average of 30 months
  The progression free survival of the enrolled patients from starting VT3989 treatment
Quality of life assessment (Part 2, expansion cohort 3, 4, and 5) | Through study completion, an average of 30 months
  Assessing the Quality of life changes via patient reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Neelesh Sharma, MD, Study Director — Vivace Therapeutics
Locations (12):
- United States (9):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Arlington, Virginia
- Australia (3):
  - Monash Health, Clayton, Victoria
  - Peter MacCullum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yap TA, Kwiatkowski DJ, Dagogo-Jack I, Offin M, Zauderer MG, Kratzke R, Desai J, Body A, Millward M, Tolcher AW, Raghav KPS, Thurston A, Post L, Dorr FA, Tang TT, Li Y, Sharma N, Kindler HL. YAP/TEAD inhibitor VT3989 in solid tumors: a phase 1/2 trial. Nat Med. 2025 Dec;31(12):4281-4290. doi: 10.1038/s41591-025-04029-3. Epub 2025 Oct 19. PMID 41111090